CLINICAL TRIAL: NCT01617694
Title: Comparison Between Remifentanil Target-controlled Infusion and Dexmedetomidine Bolus Administration for Smooth Emergence From General Sevoflurane Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2011-0181
Record Dates: First submitted 2012-06-05; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Thyroid Neoplasm
Keywords: dexmedetomidine; remifentanil; target-controlled infusion
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- group R (Experimental): continuation of remifentanil target controlled infusion (TCI) at effect-site concentration of 2 ng/ml during anesthetic recovery until extubation.
  Interventions: Drug: dexmedetomidine; Drug: Normal Saline
- group D (Active Comparator): remifentanil TCI discontinuation and dexmedetomidine 0.5 mg/kg intravenous injection before 10 min of the end of surgery
  Interventions: Drug: dexmedetomidine; Drug: Normal Saline

INTERVENTIONS:
Drug: dexmedetomidine — Fifteen minutes before the end of surgery, the first practitioner replace the syringe of remifentanil as new one; new syringe contains remifentanil in remifentanil group (Group R), and normal saline in dexmedetomidine group (Group D), respectively. There are no drug labeling in the new syringe, so the second practitioner can't know which drug was contained in the new syringe. Simultaneously, the second practitioner remifentanil concentration on monitor of TCI pump will be adjusted to 2.0 ng•ml-1. Ten minutes before the end of surgery, 10 ml of dexmedetomidine 0.5 mcg•kg-1 mixed with normal saline will be given for 5 min in Group D; in Group R, 10 ml of normal saline will be given by the first practitioner.
Drug: Normal Saline

SUMMARY:
Remifentanil target-controlled infusion and dexmedetomidine single-dose administration are known to reduce airway response and haemodynamic stimulation during anaesthetic recovery. The investigators will compare the effects of two drugs on prevention of cough during emergence from general sevoflurane anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* female patient,
* aged 20-60 yr,
* ASA physical status 1-2,
* patients undergoing elective thyroidectomy under general anesthesia

Exclusion Criteria:

* sighs of difficult airway,
* history of respiratory disease or chronic cough,
* cardiovascular disease,
* pregnant or breast-feeding woman.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
coughing response | from discontinuation of anesthetic agent (sevoflurane) to 5 min after extubation.
  Emergence cough was defined as the cough occurrence during peri-extubation period, from sevoflurane discontinuation to 5 min after extubation. The severity of cough was assessed and recorded by the following cough grading system: Grade 0, no cough; Grade 1, single cough with mild severity; Grade 2, cough persistence less than 5 s with moderate severity; Grade 3, severe, persistent cough for more than 5 s (bucking).

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Lee B, Lee JR, Na S. Targeting smooth emergence: the effect site concentration of remifentanil for preventing cough during emergence during propofol-remifentanil anaesthesia for thyroid surgery. Br J Anaesth. 2009 Jun;102(6):775-8. doi: 10.1093/bja/aep090. Epub 2009 May 2. PMID 19411668
- [Background] Guler G, Akin A, Tosun Z, Eskitascoglu E, Mizrak A, Boyaci A. Single-dose dexmedetomidine attenuates airway and circulatory reflexes during extubation. Acta Anaesthesiol Scand. 2005 Sep;49(8):1088-91. doi: 10.1111/j.1399-6576.2005.00780.x. PMID 16095449
- [Background] Turan G, Ozgultekin A, Turan C, Dincer E, Yuksel G. Advantageous effects of dexmedetomidine on haemodynamic and recovery responses during extubation for intracranial surgery. Eur J Anaesthesiol. 2008 Oct;25(10):816-20. doi: 10.1017/S0265021508004201. Epub 2008 Apr 10. PMID 18400140
- [Background] Nho JS, Lee SY, Kang JM, Kim MC, Choi YK, Shin OY, Kim DS, Kwon MI. Effects of maintaining a remifentanil infusion on the recovery profiles during emergence from anaesthesia and tracheal extubation. Br J Anaesth. 2009 Dec;103(6):817-21. doi: 10.1093/bja/aep307. Epub 2009 Oct 28. PMID 19864308